CLINICAL TRIAL: NCT02687945
Title: Study to Evaluate Outpatient Physiotherapy in Total Hip Arthroplasty: A Prospective Randomized Controlled Trial
Brief Title: PT vs no PT Following THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: 2016MAus
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (2):
- Outpatient physiotherapy (Active Comparator): two weeks of in-home physiotherapy following total hip replacement followed by two months of outpatient physiotherapy with 2-3 weekly sessions
  Interventions: Procedure: Outpatient physiotherapy
- No outpatient physiotherapy (Active Comparator): two weeks of in-home physiotherapy following total hip replacement followed by two months of self-guided physiotherapy exercises
  Interventions: Procedure: Self-guided physiotherapy

INTERVENTIONS:
Procedure: Outpatient physiotherapy
  Arms: Outpatient physiotherapy
Procedure: Self-guided physiotherapy
  Arms: No outpatient physiotherapy

SUMMARY:
The purpose of this study is to determine if outpatient physiotherapy results in improved and/or more rapid achievement of functional outcomes and quality of life in comparison to those patients who do not undergo outpatient physiotherapy after total hip arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing unilateral primary total hip arthroplasty with age > 60

Exclusion Criteria:

* Post-traumatic osteoarthritis
* Rheumatoid arthritis or other peripheral inflammatory disease
* Avascular necrosis
* Revision or conversion THA
* Post-septic osteoarthritis
* Patients discharged to a rehabilitation unit or other form of respite care such as a skilled nursing facility, acute rehabilitation center, convalescent home, long-term care facility or nursing home

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 4 weeks
  This is a validated instrument